CLINICAL TRIAL: NCT04437160
Title: A Multicenter, Randomised, Open-label Phase II Study to Evaluate the Efficacy and Safety of Adjuvant Chemotherapy for Triple Negative Breast Cancer Patients With Residual Disease After Platinum-based Neoadjuvant Chemotherapy
Brief Title: Adjuvant Chemotherapy for Triple Negative Breast Cancer Patients With Residual Disease After Neoadjuvant Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pin Zhang, Clinical Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC2019L06
Record Dates: First submitted 2020-06-05; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple negative breast cancer; Neoadjuvant chemotherapy; Residual invasive breast cancer; Adjuvant chemotherapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Epirubicin; pirarubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adjuvant chemotherapy (Experimental): Adjuvant chemotherapy for triple negative breast cancer with residual invasive disease (invasive breast tumor size≥1cm and/or positive axillary lymph nodes) after taxanes and platinum based neoadjuvant chemotherapy.
  Adjuvant chemotherapy regiments: Epirubicin 80-90mg/m2 IV or Pirarubicin 50mg/m2 IV + Cyclophosphamide 600mg/m2 IV, q21d*4cycles.
  Interventions: Drug: Epirubicin or Pirarubicin; Drug: Cyclophosphamide
- Observation (No Intervention): No adjuvant chemotherapy for triple negative breast cancer with residual invasive disease (invasive breast tumor size≥1cm and/or positive axillary lymph nodes) after taxanes and platinum based neoadjuvant chemotherapy.

INTERVENTIONS:
Drug: Epirubicin or Pirarubicin — Epirubicin 80-90mg/m2 IV or Pirarubicin 50mg/m2 IV, q21d*4cycls
  Other Names: EPI or THP
  Arms: Adjuvant chemotherapy
Drug: Cyclophosphamide — Cyclophosphamide 600mg/m2 IV, q21d*4cycls
  Other Names: CTX
  Arms: Adjuvant chemotherapy

SUMMARY:
This study will evaluate the efficacy and safety of antharcycline-based adjuvant chemotherapy compared with observation in triple negative breast cancer (TNBC) patients with residual invasive disease after platinum and taxanes based neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, phase II study. TNBC patients with residual invasive disease (invasive breast tumor size≥1cm and/or positive axillary lymph nodes) after platinum and taxanes based neoadjuvant chemotherapy are enrolled (n = 286). Patients are assigned to the chemotherapy group or the observation group at a 1:1 ratio randomly 4-6 weeks after surgery. Patients in the chemotherapy group are given anthracycline combined with cyclophosphamide regimen for 4 cycles. At the same time, the blood and tissue samples are collected for relevant tests. Follow up every 3-6 months and record recurrences and deaths.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed invasive adenocarcinoma of the breast.
* Triple negative breast cancer: hormone receptor negative (ER < 10% and PgR < 10%) and HER2 negative (IHC 0/1+ or ISH non-amplified), as defined by the local pathology laboratory.
* Clinical stage at presentation: T1-4, N0-3, M0, with indications for neoadjuvant chemotherapy.
* Patient must have received platinum and taxanes neoadjuvant chemotherapy for at least 4 cycles and no tumor progression occurred.
* Patients should have undergone adequate tumor excision in the breast and lymph nodes after neoadjuvant chemotherapy.
* Residual invasive disease must be ≥1cm in the breast, and/or have positive axillary lymph nodes observed on pathologic exam after neoadjuvant chemotherapy.
* ECOG Performance Status: 0-1.
* Patients without severe heart, lung, liver and kidney disease.
* Adequate hematologic and end-organ function.
* No more than 6 weeks may elapse between definitive breast surgery and randomization.

Exclusion Criteria:

* Previous neoadjuvant chemotherapy with anthracycline or other drugs (except platinum and taxanes).
* Previous neoadjuvant chemotherapy with platinum or taxanes alone.
* Patients have received other adjuvant therapy.
* Comprehensive medical examinations have revealed distant metastases before randomization.
* Patients who are not suitable for anthracycline evaluated by investigators.
* Prior history of other malignancy (except carcinoma in situ).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
RFS | median 5 years
  RFS defined as the time from randomization to the first recurrence event or death through the end of study

SECONDARY OUTCOMES:
OS | median 5 years
  OS defined as the time from randomization to all-cause death through the end of study
Percentage of patients with adverse events | 2-3 years
  To assess the toxicity of adjuvant chemotherapy by CTCAE v5.0
Changes in patient-reported quality of life | 2-3 years
  To assess the mean changes from baseline score in patient-reported quality of life using EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Pin ZHANG, MD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital & Institute Chinese Academy of Medical Sciences (CAMS), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No